CLINICAL TRIAL: NCT02960308
Title: A Pilot Study of Whole-Neck CT Perfusion With the Toshiba Aquilion ONE ViSION-320 Detector Row CT Scanner for Use in Head &Amp; Neck Tumor Patients
Brief Title: Whole-Neck Computed Tomography Perfusion Scan in Imaging Patients With Head and Neck Tumors
Status: Completed | Type: Observational
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 7H-16-2; NCI-2016-01583 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 7H-16-2 (Other: USC / Norris Comprehensive Cancer Center); P30CA014089 (NIH)
Record Dates: First submitted 2016-11-07; First posted 2016-11-09 (Estimated); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Head and Neck Neoplasm; Malignant Head and Neck Neoplasm
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Cytidine Triphosphate

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Diagnostic (WNCTP scan): Patients undergo WNCTP scan over 2-3 minutes during standard of care CT.
  Interventions: Radiation: Computed Tomography Perfusion Imaging

INTERVENTIONS:
Radiation: Computed Tomography Perfusion Imaging — Undergo WNCTP scan

SUMMARY:
This pilot clinical trial studies how well whole-neck computed tomography perfusion scans work in imaging patients with head and neck tumors. Diagnostic imaging procedures, such as whole-neck computed tomography perfusions scans, may provide more information about the blood supply to head and neck tumors which may help doctors plan better treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the difference in whole-neck computed tomography perfusion (WNCTP) parameters (blood volume [BV], blood flow [BF], capillary permeability [CP] and mean transit time [MTT]) between head and neck tumor masses (benign or malignant) and adjacent normal skeletal muscle within the same patient.

II. To assess whether the difference in WNCTP parameters between tumor masses and adjacent normal skeletal muscle is different between patients with benign tumor versus (vs.) malignant tumor.

III. To assess the correlation in WNCTP parameters between tumor masses and adjacent normal skeletal muscle.

IV. Determine if more suspicious cervical lymph nodes will be seen using the whole-neck coverage employed in WNCTP compared to the limited coverage of traditional neck CTP.

OUTLINE:

Patients undergo WNCTP scan over 2-3 minutes during standard of care computed tomography (CT).

After completion of study, patients are followed up within 2 days.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed or suspected head and neck tumor (benign or malignant)
* Scheduled for contrast CT (standard of care)
* No known allergies to contrast material

Exclusion Criteria:

* Known allergies to contrast material
* Pregnant or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients seen at USC/Norris Comprehensive Cancer Center who have confirmed or suspected head and neck tumor (benign or malignant) who are scheduled for contrast CT (standard of care) will be recruited for the study.
Sampling Method: Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2016-10-20 (Actual); Primary Completion 2021-06-14 (Actual); Study Completion 2021-06-14 (Actual)

PRIMARY OUTCOMES:
Number and site of each suspicious lymph node assessed by WNCTP | Day 1
  Will be compared to traditional neck CTP. Within each patient, the number and sites of each suspicious lymph node will be recorded for the whole-neck imaging area. A 95% confidence interval for the proportion of patients whose status (lymph node negative [LN-] versus lymph node positive [LN+]) was changed based on the WNCTP image compared to standard of care will be constructed.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Shiroishi, Principal Investigator — University of Southern California
Locations (1):
- USC / Norris Comprehensive Cancer Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No